CLINICAL TRIAL: NCT06140277
Title: Using Of Chitosan in Alveolar Ridge Preservation: Randomized Clinical Trial.
Brief Title: Using Of Chitosan in Alveolar Ridge Preservation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Prince Sattam Bin Abdulaziz University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PrinceSBAU
Record Dates: First submitted 2023-07-09; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Tooth Extraction Status Nos; Bone Augmentation
Keywords: chitosan; socket preservation
MeSH Terms: interventions — Bone Transplantation; Chitosan

STUDY DESIGN:
Intervention Model Description: There will be a total of 3 groups (10 patients for each), first group will be treated using chitosan as a replacement of bone particles with collagen membrane. 2nd group will be treated using the gold standard protocol which is the allograft bone particles with collagen membrane, and the last group will received nothing as control
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: For randomization, The investigator will send a form to the study therapist who is not involved in assessing outcome of the study. This form will include a randomization number. In the clinic, closed envelopes with printed randomization numbers on it are available. For every randomization number the corresponding code for the therapy group of the randomization list will be found inside the envelopes. The therapist will open the envelope and will find the treatment protocol to be conducted in this patient. Staff responsible for recruitment and outcome assessor is not allowed to receive information about the group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Chitosan (Experimental): group will be treated using chitosan as a replacement of bone particles with collagen membrane after tooth extraction
  Interventions: Procedure: extraction with chitosan particles as a replacement for bone graft with collagen membrane
- Allograft (Active Comparator): after extraction, the group will be treated using the gold standard protocol which is the (allograft) bone particles with collagen membrane.
  Interventions: Procedure: extraction with placing of allograft particles with collagen membrane
- placebo (Placebo Comparator): the extraction will be done without placing any bone material inside
  Interventions: Procedure: tooth extraction only

INTERVENTIONS:
Procedure: extraction with chitosan particles as a replacement for bone graft with collagen membrane — to replace the bone at the extraction site we will put either chitosan or allograft particles
  Other Names: chitosan
  Arms: Chitosan
Procedure: extraction with placing of allograft particles with collagen membrane — to replace the bone at the extraction site we will put allograft particles
  Other Names: gold standard treatment
  Arms: Allograft
Procedure: tooth extraction only — hopeless tooth will be extracted without any intervention
  Other Names: normal extraction
  Arms: placebo

SUMMARY:
The goal of this clinical trial is to assess the efficacy of chitosan as a socket preservation material after tooth extraction in compare to the standard treatment. The study will include patients who exhibit hopeless tooth without any periodontal infection. Smokers, history of allergy, patients with major medical issue and pregnant women will be excluded from the study. The main question[s] to answer is : is there a significant difference in bone density and dimension between the test and control groups after tooth extraction or not.

Participants will be asked to do CBCT scan and take upper and lower impressions before extraction and after three month from extraction. Then, the patients will randomly assigned to one from these groups: There will be a total of three groups (10 patients for each), first group will be treated using mixed of chitosan and allograft, second group will be treated using allograft alone and the last group will be used as control. All patients will be treated in accordance with the 2013 Declaration of Helsinki.

DETAILED DESCRIPTION:
To evaluate the tissue response, intraoral impressions and X-ray will be taking from each patient before extraction and three months after. Also, Cone-beam computed tomography (CBCT) will be taking to measure the bone growth at base line and three months after surgery is done. For measurement, each socket will be vertically divided into 3 equal areas: coronal, middle, and apical. Regenerated bone density will be assessed in each area, in both control and intervention groups.

Data then can be analyzed using SPSS ver. 11 (SPSS Inc., Chicago,USA). P-values less than 0.05 were considered as significant.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of hopeless tooth.
* Healthy patient.
* Healthy gingiva without any periodontal disease.
* Patient is welling to come after three months.

Exclusion Criteria:

* Smokers.
* History of allergy.
* pregnant women.
* patient with systemic disease.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-18 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-03-20 (Estimated)

PRIMARY OUTCOMES:
Bone Hight | 3 months
  Changes in vertical dimension in mm from baseline using scans section from CBCT.
Bone volume | 3 months
  Changes in horizontal width in mm from baseline using scans section from CBCT.

SECONDARY OUTCOMES:
Tissue healing | 3 months
  changes in scale of redness of gingiva from baseline
Dry socket | 3 months
  the No of exposed bone from baseline until healing

CONTACTS AND LOCATIONS:
Locations (1):
- Prince Sattam Bin Abdulaziz University, Riyadh, Central, Saudi Arabia